CLINICAL TRIAL: NCT05264142
Title: Impact of Genetic Polymorphism on Drug Interactions Involving CYP2C19: Risk of Phenoconversion in Healthy CYP2C19 Fast, Normal and Intermediate Metabolizers Status
Brief Title: Risk of CYP2C19 Phenoconversion in Healthy Volunteers With Rapid, Normal, and Intermediate Predicted Metabolizers' Status
Acronym: Switch19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Caroline Samer, Professor, University Hospital, Geneva
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-XXXX
Record Dates: First submitted 2022-02-11; First posted 2022-03-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Healthy
Keywords: Phenoconversion; Pharmakinetics; Genotype; Cytochrome 2C19
MeSH Terms: interventions — Voriconazole; Fluvoxamine; Tablets; Omeprazole

STUDY DESIGN:
Intervention Model Description: The study will include 3 distinct CYP2C19 genotype groups that will constitute the 3 arms of the study. For each volunteer, the study will consist of 3 sessions. Same drugs will be administered to the 3 arms of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CYP2C19 Rapid Metabolizers (RM) (Experimental): CYP2C19 rapid metabolizers (RM) are characterized by one normal function allele and one increased function allele
  Interventions: Drug: Voriconazole 200mg; Drug: FluvoxaMINE 50 Mg Oral Tablet; Drug: Omeprazole 10 MG Oral Tablet
- CYP2C19 Normal metabolizers (NM) (Experimental): CYP2C19 normal metabolizers (NMs) harboring two normal function alleles defined by the lack of any characterized polymorphisms.
  Interventions: Drug: Voriconazole 200mg; Drug: FluvoxaMINE 50 Mg Oral Tablet; Drug: Omeprazole 10 MG Oral Tablet
- CYP2C19 Intermediate metabolizers (IM) (Experimental): CYP2C19 intermediate metabolizers (IMs) are characterized by the presence of one normal function allele and one no function allele or one no function allele and one increased function allele.
  Interventions: Drug: Voriconazole 200mg; Drug: FluvoxaMINE 50 Mg Oral Tablet; Drug: Omeprazole 10 MG Oral Tablet

INTERVENTIONS:
Drug: Voriconazole 200mg — Voriconazole is a weak CYP2C19 inhibitor. It is used in study session 2 to study the impact of a weak inhibitor on the phenotype switch among the different genotypes included in the study.
  Other Names: J02AC03
Drug: FluvoxaMINE 50 Mg Oral Tablet — Fluvoxamine is a strong CYP2C19 inhibitor. It is used in study session 3 to study the impact of a strong inhibitor on the phenotype switch among the different genotypes included in the study.
  Other Names: N06AB08
Drug: Omeprazole 10 MG Oral Tablet — Omeprazole is a CYP2C19 probe substrate. It is used in the study as a tool for CYP2C19 phenotyping at each of the sessions.
  Other Names: A02BC01

SUMMARY:
CYP2C19 is responsible for the metabolism of approximately 10% of drugs currently on the market, including several proton pump inhibitors, clopidogrel, benzodiazepines and some tricyclic antidepressants, including amitriptyline. It is a cytochrome whose activity is characterized by a great variability in the general population. This variability can be explained, in part, by genetic and environmental factors The classification of phenotypes associated with CYP2C19 has evolved over time. Today, five distinct phenotypes are used to characterize this variability: the slow metabolizer (SM) phenotype, the intermediate metabolizer (IM) phenotype, the normal metabolizer (NM) phenotype, the fast metabolizer (RM) phenotype and finally the ultra-fast metabolizer (UM) phenotype. (UM) phenotype.

Although directly measurable with test substances, CYP2C19 phenotypes are often assigned on the basis of genotype. They may be impacted by intrinsic (e.g., comorbidities) or extrinsic (e.g., co-medications) factors. Phenoconversion or phenotypic change is the phenomenon by which an individual switches from one phenotype to another due to an environmental influence such as a drug interaction. However, genotype is likely to influence the degree of response to a drug interaction. Vulnerability to phenoconversion therefore differs according to the genotype of the individual.

The purpose of our study is to determine whether individuals genetically MR, NM and IM have the same vulnerability to phenoconversion. Thus, the magnitude of the response to CYP2C19 inhibition will be studied in these 3 groups of individuals (NM:*1/*1, RM:*1/*17 and IM:*1/*2-*2/*17). Inhibition will be studied in two steps, using a strong (fluvoxamine) and a weak (voriconazole) inhibitor of CYP2C19.

DETAILED DESCRIPTION:
Phase 1, open-label, parallel study in healthy volunteers selected according to their genotypic belonging to one of the three study groups.

Volunteers are included in the study and go through a buccal swab for genotyping, allowing their allocation into 3 groups according to their CYP2C19 genotype (RM: *1/*17 - NM: *1/*1 - IM: *1/*2 and *2/*17).

Following this step, volunteers have an inclusion session to determine if they meet the inclusion and non-exclusion criteria for the study.

The included volunteers will participate in three study sessions will take place.

Session 1 (control session): administration of 10mg of omeprazole for CYP2C19 phenotyping Session 2: same as session 1 with a prior intake of voriconazole 400 mg (weak inhibitor of CYP2C19 2 hours before omeprazole intake) Session 3: same as session 1 with a prior intake of fluvoxamine (strong CYP2C19 inhibitor, 12 h before and 2 h before taking the omeprazole)

At each session, dried blood spot (DBS) samples will be collected before the intake of the omeprazole (T0) and then at 2, 3, 6 and 8 hours after taking the capsule.

A wash-out period of minimum 3 days will be observed between session 1 and 2 and of minimum 1 week will be observed between sessions 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women ≥ 18 years old
* Understanding of French language and able to give a written consent
* Reliable contraception during the whole study, including a barrier method
* CYP2C19 genotype associated to the RM (*1/*17) , NM(*1/*1) AND IM(*1/*2-*2/*17) activity groups

Exclusion Criteria:

* Participation in any other interventional clinical study within 3 months prior to inclusion
* Pregnant or breastfeeding woman
* Any pathologies, use of drugs or food that may affect CYP activity (based on the "drug interactions and cytochromes P450" table published by the service of Clinical Pharmacoloy and Toxicology, HUG and on the investigator's knowledge)
* History of liver transplantation
* Alcohol intake during fluvoxamine intake
* Psychotropic substances use during fluvoxamine intake
* Alteration of hepatic tests (ASAT, ALAT, GGT, BILI) more than 3x normal
* Glomerular filtration rate (GFR) < 60 ml/min/1.73 m2
* Medical history of chronic alcoholism or abuse of psychoactive drugs
* Regular use of psychotropic substances
* Sensitivity to any of the drugs used
* Psychiatric disorders
* Beck Score ≥ 10 (question related to suicide >0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Phenoconversion rate | 2 months
  The proportion of volunteers in each group who acquire a phenotype switch such as from NM to PM after pre-treatment by voriconazole and fluvoxamine (weak and strong inhibitors, respectively)

SECONDARY OUTCOMES:
AUC assessment | 1 year
  Test drugs and their metabolite AUC measurement in whole capillary blood as well as metabolite /probe AUC ratio and single points metabolic ratios.
CL assessment | 1 year
  Test drugs and their metabolite Cl measurement in whole capillary blood
Cmax assessment | 1 year
  Test drugs and their metabolite Cmax measurement in whole capillary blood
Tmax assessment | 1 year
  Test drugs and their metabolite Tmax measurement in whole capillary blood

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Samer, Prof, Principal Investigator — Division of Clinical Pharmacology and Toxicology, Department of Anesthesiology, Pharmacology, Intensive Care and Emergency Medicine, Geneva University Hospitals
Locations (1):
- Geneva University Hospitals, HUG, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No